CLINICAL TRIAL: NCT03959228
Title: Impact of Low Protein Diet Supplemented With Ketoanalogues on Uremic Toxins Production and Glucose Metabolism in Chronic Kidney Disease
Brief Title: Impact of Low Protein Diet Supplemented With Ketoanalogues Supplementation on Uremic Toxins Production
Acronym: KETO-GUT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL18_0957
Record Dates: First submitted 2019-04-25; First posted 2019-05-22 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- referencial diet (No Intervention): 0.8 g/kg/day of protein
- protein very poor diet with additional keto-analogs (Experimental): 0.4 g/kg/day of protein and 1 pill of Ketosteril/ 5kg.
  Interventions: Drug: keto-analogs

INTERVENTIONS:
Drug: keto-analogs — The patients that will be included in the experimental arm will have additional keto-analogs (1 pill/5 kg).
  Arms: protein very poor diet with additional keto-analogs

SUMMARY:
Chronic kidney disease (CKD) is associated with accumulation of uremic toxins like p-cresyl sulfate and indoxyl sulfate that are associated of cardiovascular complication and perturbation of glucose metabolism. These toxins are produced by fermentation of protein by intestinal microbiota but the role of low protein diet and ketoanalogue supplementation on uremic toxins production and microbiota composition are unknown. Low protein diet supplemented with ketoanalogues is recommended inCKD patients to prevent progression of renal disease. The aim of this study is to determine the impact of uremic toxins concentration, microbiota composition and gut hormone involved in carbohydrate metabolism ( GLP-1, FGF19, bile acids) with low protein diet supplemented with ketoanalogues.

ELIGIBILITY:
Inclusion Criteria:

* CKD stage 4-5 with estimated glomerular filtration rate < 30 ml/min/1,73m2
* No dialysis
* No history of kidney transplantation
* Non-diabetic (fasting glucose <1.26 g / L, or no insulin or oral antidiabetic therapy)
* BMI between 18 and 30 kg / m2
* Patient followed in the nephrology department of Professor FOUQUE at the Lyon Sud hospital
* For women of childbearing age, at least one method of contraception recognized as effective
* Patient who gave consent to open participation and signed the consent to participate in the study

Exclusion Criteria:

* Patient with progressive inflammatory, infectious, cardiovascular or neoplastic disease
* Patient refusing a dietary follow-up
* Patient having a planned transplant or dialysis project in the next 6 months.
* Patient having a colectomy, resection of the small intestine or cholecystectomy
* Patient who has received antibiotics, prebiotics, probiotics in the last 3 months.
* Patient treated with more than 2 g of calcium per day
* Patient using laxatives (more than 2 per day)
* Patient having:
* Uncontrolled metabolic acidosis (bicarbonatemia <18 mM)
* Hyperparathyroidism (PTH greater than 5 times the upper limit of normal)
* Hypercalcemia (Calcium> 2.55 mmol / L) or hypophosphoremia <0.70 mmol / L
* Anemia (hemoglobinemia <80g / L)
* Undernutrition criteria: albumin <38 g / L or prealbumin <0.3 g / L
* Known hypersensitivity to any of the substances or excipients of Ketosteril
* Subject in exclusion period of a previous study
* Patient not affiliated to social security
* Patient under guardianship or in the interests of justice
* Patient who is pregnant, breastfeeding or likely to become pregnant during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-11-12 (Actual); Primary Completion 2023-12-12 (Estimated); Study Completion 2023-12-12 (Estimated)

PRIMARY OUTCOMES:
Indoxyl Sulfate Plasmatic concentration | After 3 months of diet
  Concentration mesure of Indoxyl Sulfate Plasmatic

SECONDARY OUTCOMES:
TMAO uremic toxin concentraction ( TMAO, PCS) in plasma | After 3 months
  concentration mesure of uremic toxin in plasma
TMAO uremic toxin concentraction in urine ( IS, PCS) | After 3 months
  concentration mesure of uremic toxin in urine
Composition of intestinal microbiota | Before three months
  sequencing 16s stool samples
Composition of intestinal microbiota | After three months
  sequencing 16s stool samples
Insulin sensitivity | After 3 months
  oral glucose tolerance test
Insulin secretion | After 3 months
  oral glucose tolerance test
Secretion of gut hormone like GLP-1 and FGF19 | After 3 months
  oral glucose tolerance test
Composition of bile acid | After 3 months
  composition of bile acid mesure by chromatography
Concentration of bile acid | After 3 months
  concentration of bile acid mesure by Chromatography
Concentration of endotoxinemia (LPS) | After 3 months
  LPS concentration mesure
Nutritional status | After 3 months
  Nutrional status will be determined with body weight, body composition with bioimpedecemetry, albumin, prealbumin, muscle status with hand grip.
Calcemia | After 3 months
  calcemia mesure
Observance of diet | After 3 months
  counting of returned ketosteril tablets

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Lyon SUD, Pierre-Bénite, France